CLINICAL TRIAL: NCT06252480
Title: Effect of Various Intensities of tDCS on Dual Task Cognitive Functions in Normal Subjects: A Pilot Study
Brief Title: Effect of Various Intensities of tDCS on Dual Task Cognitive Functions in Normal Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Subhasish Chatterjee, Effect of various intensities of tDCS on dual task cognitive functions in normal subjects: A Pilot Study, Maharishi Markendeswar University (Deemed to be University)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPC-PA-07
Record Dates: First submitted 2024-02-02; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Functions
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensities of tDCS and dual task cognitive functions (Experimental): We have done in a one arm type. The participants are divided into different intensity group (0.5 mA, 1.0 mA, 1.5 mA and 2.0 mA).
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — 4 variance of different intensities of tDCS (0.5mA, 1 mA, 1.5mA and 2mA). At F3 and F4, tDCS was applied to the desired region. Electrodes were put in using the 10-20 EEG technique throughout the parietal cortex, with the current electrode being set on F3 area and control electrode being positioned on the F4 area. For 20 minutes over three days per week for up to three weeks, current intensities of 0.5mA for group A, 1.0mA for group B, 1.5mA for group C, and 2.0mA for group D were administered. when engaging in dual-task cognitive processes. The groups are going to receive 9 sessions of tDCS treatment.

SUMMARY:
Transcranial Direct Current Stimulation (tDCS) is a neuroregulatory method that delivers a weak straight tendency to neuronal areas with the intention of changing the brain's basic metabolic processes. Degradation of executive performance may not necessarily arise from cathodal stimulation, and vice versa for anodal stimulation.

DETAILED DESCRIPTION:
Total 48 samples were taken, were randomly allocated into an experimental group of 4 variance of different intensities of tDCS. At F3 and F4, tDCS was applied to the desired region. Electrodes were put in using the 10-20 EEG technique throughout the parietal cortex, with the current electrode being set on F3 area and control electrode being positioned on the F4 area. For 20 minutes over three days per week for up to three weeks, current intensities of 0.5mA for group A, 1.0mA for group B, 1.5mA for group C, and 2.0mA for group D were administered. when engaging in dual-task cognitive processes. The groups are going to receive 9 sessions of tDCS treatment. The MoCA and TMT scale was completed by samples before and after the intervention. Finally, specifics investigation will be carried out using SPSS 26.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy students only
* Willing to participate in the study

Exclusion Criteria:

* Any recent trauma or injury on the head of subjects
* If contact with the scalp is not possible
* Any resonant implant close to electrode placement site

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
MoCA | 10 mins
  A quick test for minor cognitive impairment. It evaluates a variety of cognitive processes, including executive functioning, recall, speech and direction. The assessment has 30 points and requires 10 mins to finish for each person. A typical result is that 26 and more is normal.

SECONDARY OUTCOMES:
TRAIL MAKING TEST | 3 minutes
  TMT part A includes 25 rounds containing the digits 1 to 25 scribbled haphazardly within every round on a sheet of paper. TMT part B similarly includes 25 rounds on a sheet of paper, but this rounds includes digits (1-12) and alphabet (A-L) instead of only being digits.

CONTACTS AND LOCATIONS:
Overall Officials: Subhashish Chatterjee, MPT(NEURO), Principal Investigator — Maharishi Markendeshwar Institute of Physiotherapy and Rehabilitation, Ambala, Haryana, 133207
Locations (1):
- MMIPR, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No